CLINICAL TRIAL: NCT05239143
Title: A Phase 1 Dose Escalation and Expanded Cohort Study of P-MUC1C-ALLO1 in Adult Subjects With Advanced or Metastatic Solid Tumors
Brief Title: P-MUC1C-ALLO1 Allogeneic CAR-T Cells in the Treatment of Subjects With Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Poseida Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P-MUC1C-ALLO1-001
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Ovarian Cancer; Non Small Cell Lung Cancer; Colorectal Cancer; Pancreatic Cancer; Renal Cell Carcinoma; Nasopharyngeal Cancer; Head and Neck Squamous Cell Carcinoma; Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Renal Cell; Nasopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, 3 + 3 design of dose-escalating cohorts with open label, dose expansion at recommended phase 2 dose (RP2D)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- P-MUC1C-ALLO1 CAR-T cells (Single Dose - Arm A) (Experimental): * Single ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following lymphodepletion regimen 1.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid
- P-MUC1C-ALLO1 CAR-T cells (Multiple Dose - Arm B) (Experimental): * Cyclic administration of ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following lymphodepletion regimen 1.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid
- P-MUC1C-ALLO1 CAR-T cells (Single Dose - Arm C) (Experimental): * Single ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following lymphodepletion regimen 2.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid
- P-MUC1C-ALLO1 CAR-T cells (Multiple Dose - Arm D) (Experimental): * Cyclic administration of ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following lymphodepletion regimen 2.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid
- P-MUC1C-ALLO1 CAR-T cells (Single Dose - Arm A1) (Experimental): * Single ascending A1 dose cohorts, given in a single intravenous infusion of CAR-T cells, following lymphodepletion regimen 1.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid
- P-MUC1C-ALLO1 CAR-T cells (Single Dose - Arm E) (Experimental): * Single ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following assigned lymphodepletion regimen.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid
- P-MUC1C-ALLO1 CAR-T cells (Multiple Dose - Arm F) (Experimental): * Cyclic administration of ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following assigned lymphodepletion regimen.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid
- P-MUC1C-ALLO1 CAR-T cells (Single Dose - Arm M) (Experimental): * Single ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following assigned lymphodepletion regimen.
  * Rimiducid may be administered as indicated.
  Interventions: Biological: P-MUC1C-ALLO1 CAR-T cells; Drug: Rimiducid

INTERVENTIONS:
Biological: P-MUC1C-ALLO1 CAR-T cells — P-MUC1C-ALLO1 is an allogeneic CAR-T cell therapy designed to target cancer cells expressing MUC1-C.
Drug: Rimiducid — Rimiducid (safety switch activator) may be administered as indicated.

SUMMARY:
A Phase 1, open label, dose escalation and expanded cohort study of P-MUC1C-ALLO1 in adult subjects with advanced or metastatic epithelial derived solid tumors, including but not limited to the tumor types listed below.

DETAILED DESCRIPTION:
This is an open label, multi-center Phase 1 study that will follow a 3 + 3 design of dose-escalating cohorts of single and multiple doses of P-MUC1C-ALLO1 to determine a Recommended Phase 2 Dose (RP2D). P-MUC1C-ALLO1 is an allogeneic chimeric antigen receptor (CAR) T cell therapy designed to target cancer cells expressing Mucin1 cell surface associated C-Terminal (MUC1-C) antigen. Additional participants will be treated with P-MUC1C-ALLO1 at the determined RP2D.

Following enrollment, subjects will be treated with P-MUC1C-ALLO1 and will undergo serial measurements of safety, tolerability and response. Rimiducid may be administered as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, Subjects ≥18 years with life expectancy >3 months
* Must have a confirmed diagnosis of unresectable, locally advanced or metastatic epithelial-derived cancer
* Must have progressed during or after last therapy, developed intolerance/toxicity to current treatment, or ineligible or refused other existing treatment options, and have measurable disease
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 or Karnofsky performance status ≥70%
* Must have adequate vital organ function within pre-determined parameters
* Must have archived tumor tissue available or consent to a biopsy collection
* Must be willing to practice birth control
* Must have a negative pregnancy test at screening and prior to initiating lymphodepletion chemotherapy or study drug administration
* Must have recovered from toxicities due to prior therapies

Exclusion Criteria:

* Has inadequate venous access
* Has an active second malignancy (not disease free for at least 5 years) in addition to the studied malignancy, excluding low-risk neoplasms such as non-metastatic basal cell or squamous cell skin carcinoma
* Is pregnant or lactating
* Has a history of or active autoimmune disease
* Has a history of significant central nervous system (CNS) disease, such as stroke, epilepsy
* Has an active systemic (viral, bacterial, or fungal) infection
* Has New York Heart Association (NYHA) Class III or IV heart failure, unstable angina, or a history of myocardial infarction or significant arrhythmia
* Has any psychiatric or medical disorder that would preclude safe participation in and/or adherence to the protocol
* Has received anticancer medications within 2 weeks of the time of initiating lymphodepletion
* Has received immunosuppressive medications within 2 weeks of administration of P-MUC1C-ALLO1, and/or expected to require them while enrolled in the study
* Has received systemic corticosteroid therapy within 1 week of the administration of P-MUC1C-ALLO1 or is expected to require it during the course of the study
* Has known CNS metastases or symptomatic CNS involvement
* Has a history of significant liver disease or active liver disease
* Has a history of known genetic predisposition to HLH/MAS
* Has received anti-cancer monoclonal antibody therapy within 4 weeks of initiating LD therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2039-04 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of P-MUC1C-ALLO1 | Baseline through Day 28
  Number of subjects with a dose limiting toxicity (DLT)
Evaluate the overall safety and tolerability profile of P-MUC1C-ALLO1 | Baseline through 15 years
  Frequency and severity of adverse events
Evaluate the preliminary efficacy of P-MUC1C-ALLO1 | Baseline through 15 years
  According to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, secondarily Immune Response Evaluation Criteria in Solid Tumors (iRECIST): Overall Response Rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Heidegger, M.D., Study Director — Lead Medical Director, Oncology, Genentech Research Early Development
Locations (14):
- United States (14):
  - University of California, Irvine Medical Center, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Maryland Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562